CLINICAL TRIAL: NCT02400671
Title: Evaluation of Mhealth Strategies to Optimize Adherence and Efficacy of PMTCT/ART
Brief Title: Mobile Strategies for Women's and Children's Health: Optimizing Adherence and Efficacy of PMTCT/ART
Acronym: Mobile WAChx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Nairobi (Other); Kenyatta National Hospital (Other Government)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000916
Record Dates: First submitted 2015-03-02; First posted 2015-03-27 (Estimated); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: mHealth; PMTCT; Adherence, Medication; SMS; Maternal Health; HIV/AIDS
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Two-way SMS (Experimental): Participants will receive weekly push SMS messaging with a questions and have the ability to text back to the study nurse
  Interventions: Behavioral: SMS messaging
- One-Way SMS (Experimental): Participants will receive weekly push SMS messaging
  Interventions: Behavioral: SMS messaging
- Control (No Intervention): Participants will receive standard of care (no intervention)

INTERVENTIONS:
Behavioral: SMS messaging
  Arms: One-Way SMS; Two-way SMS

SUMMARY:
The investigators are conducting a 3-arm randomized trial comparing the effects of unidirectional SMS (ie: "push" messaging to participant) vs. bidirectional SMS dialogue between participant and provider vs. control (no SMS) among HIV-infected Kenyan mothers in Kenyan PMTCT-ART for outcomes of ART adherence and retention in care.

DETAILED DESCRIPTION:
The investigators will compare trial arms for impact on maternal retention, adherence, virologic failure and resistance and infant HIV or HIV-free survival.

The investigators will determine correlates of maternal loss to follow-up and virologic failure and correlates of infant HIV in the overall study and stratified by trial arm. In the bidirectional SMS arm, the investigators will determine the rate of SMS interactivity, impact of critical time-points on messaging, and characteristics of high and low 'interactors'.

The investigators will determine cost-effectiveness of unidirectional and bidirectional SMS interventions. These data will contribute a potential scale-able strategy to improve PMTCT-ART as programs aspire to 'virtual elimination' of infant HIV.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, HIV-infected, access to a mobile phone, remaining in study area for two years

Exclusion Criteria:

* enrolled in another research study

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John-Stewart, Principal Investigator — UW
Locations (6):
- Kenya (6):
  - Ahero District Hospital, Ahero
  - Bondo District Hospital, Bondo
  - Mathare City Council Clinic, Nairobi
  - Riruta Health Centre, Nairobi
  - Rachuonyo sub-County Hospital, Oyugis
  - Siaya County Referral Hospital, Siaya

REFERENCES:
- [Background] Drake AL, Unger JA, Ronen K, Matemo D, Perrier T, DeRenzi B, Richardson BA, Kinuthia J, John-Stewart G. Evaluation of mHealth strategies to optimize adherence and efficacy of Option B+ prevention of mother-to-child HIV transmission: Rationale, design and methods of a 3-armed randomized controlled trial. Contemp Clin Trials. 2017 Jun;57:44-50. doi: 10.1016/j.cct.2017.03.007. Epub 2017 Mar 14. PMID 28315480
- [Background] Ronen K, Unger JA, Drake AL, Perrier T, Akinyi P, Osborn L, Matemo D, O'Malley G, Kinuthia J, John-Stewart G. SMS messaging to improve ART adherence: perspectives of pregnant HIV-infected women in Kenya on HIV-related message content. AIDS Care. 2018 Apr;30(4):500-505. doi: 10.1080/09540121.2017.1417971. Epub 2017 Dec 18. PMID 29254362
- [Background] Lewis K, Harrington EK, Matemo D, Drake AL, Ronen K, O'Malley G, Kinuthia J, John-Stewart G, Unger JA. Utilizing perspectives from HIV-infected women, male partners and healthcare providers to design family planning SMS in Kenya: a qualitative study. BMC Health Serv Res. 2019 Nov 21;19(1):870. doi: 10.1186/s12913-019-4708-7. PMID 31752872
- [Background] Fairbanks J, Beima-Sofie K, Akinyi P, Matemo D, Unger JA, Kinuthia J, O'Malley G, Drake AL, John-Stewart G, Ronen K. You Will Know That Despite Being HIV Positive You Are Not Alone: Qualitative Study to Inform Content of a Text Messaging Intervention to Improve Prevention of Mother-to-Child HIV Transmission. JMIR Mhealth Uhealth. 2018 Jul 19;6(7):e10671. doi: 10.2196/10671. PMID 30026177
- [Derived] Osborn L, Ronen K, Larsen AM, Richardson B, Khasimwa B, Chohan B, Matemo D, Unger J, Drake AL, Kinuthia J, John-Stewart G. Antenatal depressive symptoms in Kenyan women living with HIV: contributions of recent HIV diagnosis, stigma, and partner violence. AIDS Care. 2022 Jan;34(1):69-77. doi: 10.1080/09540121.2021.1981216. Epub 2021 Sep 27. PMID 34579601
- [Derived] Kinuthia J, Ronen K, Unger JA, Jiang W, Matemo D, Perrier T, Osborn L, Chohan BH, Drake AL, Richardson BA, John-Stewart G. SMS messaging to improve retention and viral suppression in prevention of mother-to-child HIV transmission (PMTCT) programs in Kenya: A 3-arm randomized clinical trial. PLoS Med. 2021 May 24;18(5):e1003650. doi: 10.1371/journal.pmed.1003650. eCollection 2021 May. PMID 34029338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 22, 2015 and May 4, 2017, participants were recruited from 6 public maternal child health (MCH) clinics in Kenya: 2 in peri-urban Nairobi County and 4 in rural Siaya, Kisumu, and Homa Bay Counties
Pre-assignment Details: 825 participants were enrolled but it was later identified that one participant was enrolled twice. Only one of these records is included in analysis for a total participant number of 824
Period: Overall Study
Arm/Group | Two-way SMS | One-Way SMS | Control
Started | 276 | 271 | 277
Completed | 249 | 239 | 249
Not Completed | 27 | 32 | 28
Not completed — Death | 5 | 3 | 4
Not completed — Lost to Follow-up | 20 | 27 | 24
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Two-way SMS: Participants will receive weekly push SMS messaging with a questions and have the ability to text back to the study nurse
  SMS messaging
- One-Way SMS: Participants will receive weekly push SMS messaging
  SMS messaging
- Total: Total of all reporting groups
Arm/Group | Two-way SMS | One-Way SMS | Control | Total
Number analyzed (Participants) | 276 | 271 | 277 | 824
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [23 to 31] | 28 [23 to 30] | 27 [23 to 31] | 27 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 271 | 277 | 824
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 276 | 271 | 277 | 824
On antiretroviral therapy (ART) >=4 months [Count of Participants; unit: Participants] | 160 | 161 | 149 | 470
Viral load (VL) >=1000 at enrollment [Count of Participants; unit: Participants] | 88 | 75 | 81 | 244
Shares phone [Count of Participants; unit: Participants] | 81 | 77 | 87 | 245
Employed [Count of Participants; unit: Participants] — Population: Missing responses
  Participants
    number analyzed (Participants) | 275 | 271 | 276 | 822
    (all) | 133 | 126 | 159 | 418
Primigravida [Count of Participants; unit: Participants] | 49 | 40 | 26 | 115

OUTCOME MEASURES:

1. Primary Outcome: Maternal Virologic Failure
Description: Prevalence of virologic failure (HIV RNA ≥1000 c/ml) after the first 4 months post-ART will be compared between study arms using Generalized Estimating Equations (GEE) with log-binomial link.
Time Frame: 2 years postpartum
Population: Participants with VL data available >=4 months post-ART initiation
Measure: Count of Units; unit: VL measurements
Units Other Than Participants: VL measurements
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 249 | 235 | 243
Number analyzed (VL measurements) | 1055 | 1066 | 1029
VL measurements | 90 | 119 | 99

2. Primary Outcome: Retention in Care
Description: Timely clinic visit attendance during follow-up from enrollment in pregnancy to 12 and 24 months postpartum will be compared between study arms using GEE with log-binomial link.
Time Frame: Assessed at 24 months postpartum
Population: Participants with clinic visits scheduled during the study period
Measure: Count of Units; unit: Scheduled visits
Units Other Than Participants: Scheduled visits
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 262 | 264 | 268
Number analyzed (Scheduled visits) | 4114 | 4124 | 4199
Scheduled visits | 3664 | 3633 | 3709

3. Primary Outcome: Loss to Follow-up
Description: The proportions of women lost to follow-up at 12 and 24 months postpartum will be compared between study arms by log-binomial regression.
Time Frame: Assessed at 24 months postpartum
Population: Participants still enrolled in the study at 24 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 267 | 270 | 276
Participants | 63 | 62 | 58

4. Primary Outcome: Infant HIV-free Survival
Description: Incidence of infant HIV acquisition or death (events per person-time of follow-up) will be compared between study arms using Cox proportional hazards regression.
Time Frame: 2 years postpartum
Population: Participants with live-born infants
Measure: Number; unit: Events
Units Other Than Participants: Person-years
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 252 | 240 | 252
Number analyzed (Person-years) | 483 | 476 | 502
Events | 20 | 11 | 13

5. Secondary Outcome: Maternal ART Adherence
Description: ART adherence, defined as the proportion of days "covered" by ART between pharmacy refills, will be dichotomized and compared between arms using GEE with log-binomial link.
Time Frame: 2 years postpartum
Population: Participants with pharmacy refill data available
Measure: Count of Units; unit: Refill visits
Units Other Than Participants: Refill visits
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 252 | 250 | 256
Number analyzed (Refill visits) | 4108 | 4096 | 4191
Refill visits | 2925 | 2881 | 2953

6. Secondary Outcome: Maternal ART Resistance
Description: Incidence of drug resistance on ART will be compared between study arms using Cox proportional hazards regression.
Time Frame: 2 years postpartum
Population: Participants without ART resistance at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Two-way SMS | One-Way SMS | Control
Number analyzed (Participants) | 246 | 248 | 254
Participants | 4 | 11 | 9

7. Secondary Outcome: Maternal Perceptions of Intervention and Care Received
Description: Qualitative interviews at exit
Time Frame: 2 years postpartum
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Pregnancy until 2 years postpartum visit (period of study enrollment)
Arm/Group | Two-way SMS | One-Way SMS | Control
All-Cause Mortality (participants affected / at risk) | 5/276 | 3/271 | 4/277
Serious Adverse Events (participants affected / at risk) | 32/276 | 18/271 | 24/277
Other Adverse Events (participants affected / at risk) | 15/276 | 17/271 | 14/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Two-way SMS (N=276) | One-Way SMS (N=271) | Control (N=277)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 5 | 3 | 4
Infant death (Pregnancy, puerperium and perinatal conditions) | 16 | 10 | 13
Maternal hospitalization (General disorders) | 5 | 1 | 3
Infant hospitalization (General disorders) | 6 | 4 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Two-way SMS (N=276) | One-Way SMS (N=271) | Control (N=277)
Miscarriage/stillbirth (Pregnancy, puerperium and perinatal conditions) | 14 | 15 | 14
Physical or sexual abuse (Social circumstances) | 0 | 2 | 0
Psychological distress (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02400671/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02400671/SAP_001.pdf
  • Informed Consent Form (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT02400671/ICF_002.pdf